CLINICAL TRIAL: NCT06995560
Title: Preliminary Investigations of Transcranial Electrical Stimulation Effects on Neurophysiology and Behavior
Brief Title: Effects of Transcranial Electrical Stimulation on Task Performance in Healthy Adults
Acronym: BRAIN-STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gary E. Strangman, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020P002253; NNX16AO30G (Other Grant/Funding Number: National Aeronautics and Space Administration (NASA))
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Brain Stimulation; Transcranial Direct Current Stimulation (tDCS); Cognition; Psychomotor Performance; Neurophysiology
Keywords: Transcranial Electrical Stimulation; Non-Invasive Brain Stimulation; Neuromodulation; Sham-Controlled Study; Double-Blind Study; Cognitive Enhancement; Working Memory; Attention; Learning and Memory; Task Performance; Human Performance; Operational Performance; Neurocognitive Function; Brain-Behavior Relationships; Dorsolateral Prefrontal Cortex; Anterior Insula; Neuronal Excitability; Functional Near-Infrared Spectroscopy (fNIRS)

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two stimulation location groups: (1) left dorsolateral prefrontal cortex (DLPFC) or (2) left anterior insula (L-aINS). Randomization is valances based on gender, age, and video gaming experience. Within each group, participants undergo a crossover design in which they receive both active and sham transcranial electrical stimulation (tES) in randomized order. This design allows for within-subject comparisons between stimulation conditions while assessing the impact of stimulation site on task performance.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators were blinded to stimulation conditions (active vs. sham) and to which pre-programmed stimulation protocol (A or B) corresponded to active stimulation. The investigator was aware of the assigned stimulation location (DLPFC or L-aINS), but not whether stimulation protocol A or B was active or sham. The tES device was operated in double-blind model, with stimulation order randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- DLPFC Stimulation Group (Experimental): Participants receive transcranial electrical stimulation (tES) targeting the left dorsolateral prefrontal cortex (DLPFC) and perform a complex cognitive-motor task using the Robotic On-Board Trainer for Research (ROBoT-r) under both active and sham stimulation in a randomized, crossover design.
  Interventions: Device: Active Transcranial Electrical Stimulation; Device: Sham Transcranial Electrical Stimulation
- Anterior Insula Stimulation Group (Experimental): Participants receive transcranial electrical stimulation (tES) targeting the left anterior insula and perform a complex cognitive-motor task using the Robotic On-Board Trainer for Research (ROBoT-r) under both active and sham stimulation in a randomized, crossover design.
  Interventions: Device: Active Transcranial Electrical Stimulation; Device: Sham Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Active Transcranial Electrical Stimulation — Active tES delivered using the Soterix Medical MXN-33 HD-tES stimulator. Stimulation is applied via high definition electrodes targeting either the left DLPFC or L-aINS at intensities up to 1.9 mA. Stimulation is performed for up to 45 minutes during task execution. Participants perform the ROBoT-r task during stimulation.
Device: Sham Transcranial Electrical Stimulation — Sham tES using the same Soterix Medical MXN-33 HD-tES stimulator and electrode placements. Stimulation ramps up and down over 20 seconds to mimic sensation but provides no continuous current. Participants perform the ROBoT-R task under sham conditions.

SUMMARY:
The objective of this randomized, double-blind, sham-controlled, crossover study is to evaluate the effects of transcranial electrical stimulation (tES) on complex cognitive task performance in healthy adult volunteers.

The primary questions this study aims to answer are:

1. Does tES improve task performance, including speed, accuracy, and overall success, during a computerized track-and-capture task?
2. Do different stimulation targets produce differential effects on performance?
3. Are there short-term post-stimulation effects on task performance (up to 48 hours)?

Participants will:

1. Complete two testing sessions under either active or sham stimulation conditions.
2. Perform a complex operational task involving dual-hand controllers while undergoing tES or sham stimulation, and immediately after.
3. Return for follow-up task performance assessments at 24 and 48 hours post-stimulation to evaluate after-effects.

DETAILED DESCRIPTION:
Transcranial electrical stimulation (tES) is a non-invasive neuromodulation technique that delivers low-intensity electrical currents (e.g., <2 mA) through scalp electrodes to modulate brain activity. Numerous studies have shown that tES can enhance cognitive functions such as learning, memory, attention, and decision-making in healthy individuals, as well as provide therapeutic benefits in psychiatric and neurological populations. Despite these findings, substantial knowledge gaps remain regarding the effects of tES, particularly in the context of complex, operationally relevant tasks.

Existing research has primarily focused on the effects of tES on simple cognitive tasks, with limited investigation into task that require multiple cognitive domain to operate simultaneously. Performance on complex tasks, such as those involving motor coordination, visual-spatial process, decision-making, and rapid response, may respond differently to tES than simple, isolated tasks. Understanding these effects could have broad applications in optimizing cognitive performance across various high-demand settings.

This study is designed to address several key uncertainties:

1. Inter-individual variability in behavioral and neurophysiological responses to tES.
2. the impact of stimulation parameters (location, type, intensity) on task performance.
3. The magnitude and duration of both immediate and post-stimulation effects on behavior.

To investigate these questions, healthy adults perform a computerized track-and-capture task requiring real-time motor control and decision-making using dual-hand controllers. Participants undergo both active and sham stimulation in a randomized, double-blind, crossover design. Stimulation will target either the left dorsolateral prefrontal cortex or the left anterior insula, guided by current flow modeling software. Performance is assessed during stimulation, immediately after, and at 24 and 48 hours post-stimulation to evaluate both immediate and short-term after-effects.

Outcome measures include task performance metrics (e.g., speed, accuracy, overall success) and neurophysiological data collected via non-invasive monitoring with functional near-infrared spectroscopy (fNIRS). The study is part of a broader research effort to characterize the functional impact of tES on complex behavior and to inform future applications in cognitive performance enhancement.

All stimulation procedures follow established safety guidelines for low-intensity tES, including continuous monitoring of electrode impedance and post-session adverse event questionnaires assessing discomfort, mood, and cognitive status. The Soterix Medical MXN-33 HD-tES system includes built-in safeguards to prevent excessive current delivery and to ensure safe electrode contact throughout the stimulation. Participants serve as their own controls in a within-subject crossover design, increasing statistical power for detecting within-subject differences between active and sham conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 55 years
* Master's or Doctorate degree, or equivalent relevant experience
* No history of head injury or neurological or psychiatric disorders
* No history of cardiac disease
* No metal implants in the head
* No implanted electronic devices
* Not taking medication affecting neural or cardiovascular function
* Able to provide written, dated informed consent

Exclusion Criteria:

* Smoking within the past year
* Current illegal drug use
* Alcohol abuse
* Pregnancy (confirmed by urine test)
* Participation in another brain stimulation protocol withing the past month

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
ROBoT-r Task Performance Score (During Stimulation) | 5 minutes after stimulation onset
  Performance on a computerized track-and-capture task assessed via a weighted score combining accuracy, speed, and success rate. Participants use dual-hand controllers to grapple a simulated spacecraft in a time-limited, physics-enabled environment. Scores from 0 to 10, with higher scores indicating better performance. Task begins 5 minutes after stimulation onset.
ROBoT-r Task Performance Score (Post-Stimulation) | 15 minutes post stimulation
  Performance On ROBoT-r task 15 minutes post-stimulation. Scored using the same weighted score (0 to 10) combining accuracy, speed, and success rate.
ROBoT-r Task Performance Score (Post-Stimulation Follow-up) | 24 and 48 hours post-stimulation
  Performance on ROBoT-r task at 24 and 48 hours post-stimulation to assess short-term after-effects. Scored using the same weighted score (0 to 10) combining accuracy, speed, and success rate.

SECONDARY OUTCOMES:
tES Adverse Effects Questionnaire | Immediately after each stimulation session
  Self-reported adverse effects following tES session, including measures of tingling, headache, fatigue, mood changes, and skin irritation. Participants rate presence and severity of effects using standardized questionnaire.
Hemodynamic Activation (HbD) - fNIRS | Post stimulation/sham and during post-stimulation session (24 and 48 hours)
  Hemodynamic brain activity measured using functional near-infrared spectroscopy (fNIRS) via the NINscan system, which was designed and built at Massachusetts General Hospital for research purposes. The NINscan system uses four dual-wavelength laser diode sources (780 nm, 830 nm) and eight photodiode detectors sampled at 250 Hz, with a 64-channel source-detector configuration. Selected channels for analysis include the left lateral, medial, and right lateral regions of the prefrontal cortex. Hemodynamic activation indexed by HbD (ΔO2Hb - ΔHHb) concentration, reflecting changes in cortical oxygenation associated with neural activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Research Institute, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD from this project will be anonymized IPD and shared. Data will be coded with a key only available to the Principal Investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available by the end-date of the funded project (estimated 12/25/2025) and retained indefinitely.
Access Criteria: Researchers will be allowed to request the data form the NASA NLSP through their website https://nlsp.nasa.gov/explore/page/home. NASA will be responsible for vetting requests and providing the data as requested.
URL: https://nlsp.nasa.gov/explore/page/home